CLINICAL TRIAL: NCT00953290
Title: Cutera Radio Frequency Device for Thigh Circumference Reduction
Brief Title: Thigh Circumference Reduction Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because the preliminary data did not indicate efficacy.
Sponsor: Cutera Inc. (Industry)
Responsible Party: Stephanie Buech, Director of Clinical Research, Cutera Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTCS002
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Reduction of Localized Excess Fat
Keywords: Cellulite; Adipose tissue; Circumference; Reduction; Thigh
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treated Thigh (Experimental): The thigh treated with the RF device
  Interventions: Device: Cutera Radio Frequency Device
- Untreated Thigh (No Intervention): The untreated thigh

INTERVENTIONS:
Device: Cutera Radio Frequency Device — Up to three treatments, one pass, dosage range of 15-60 kJ.
  Other Names: Callisto, TruForm, TruSculpt
  Arms: Treated Thigh

SUMMARY:
The purpose of this study is to evaluate the Cutera radio frequency (RF) device for the new indication of reduction of thigh circumference.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the Cutera radio frequency device for the new indication of reduction of thigh circumference.

At investigator's discretion, each subject will receive up to three treatments on one thigh and will be scheduled for two follow-up visits after the final treatment. The treated thigh will be clinically evaluated for side effects and both treated and untreated control thigh will be measured and photographed at each visit for analysis. Subjects will also be weighted at each visit and asked to fill out a survey during follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 20 and 35
* Presence of cellulite grades II, III or IV according to GLD scale
* Visible bi-lateral thigh fat Thigh area to be treated to measure at least 30.0mm in vertical fold, as measured with industry standard fat caliper
* Subject must be able to read, understand and sign the Consent Form
* Subject must adhere to the follow-up schedule and study instructions
* Subject must adhere to the same diet and/or exercise routine throughout the study

Exclusion Criteria:

* Significant weight fluctuation (+/-10 lbs) in the past 6 months
* Taking weight-loss medications/supplements
* Participation in any other clinical study
* Cellulite treatment within 3 months of the treatment
* Surgical or non-surgical treatments to the target area in the last 12 months, e.g., liposuction
* Prior treatment to the target area within the last 12 months
* Arteriosclerosis or weakened blood vessels
* Heart disease
* Thromboembolic disease
* Diagnosed or documented immune system disorders
* Bleeding disorders.
* Presence of uncontrolled hypertension
* Taking prescription anticoagulants
* History of keloid formation
* Malignant tumors in the target area
* Diabetes
* Any disease or condition that could impair wound healing
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars
* Infection in the target area
* Implanted electrical device(s)
* Pregnant or lactating

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J. Ronan, MD, Principal Investigator; Jacqueline Calkin, MD, Principal Investigator; Christine Lee, MD, Principal Investigator; Scott Kramer, MD, Principal Investigator
Locations (1):
- Blackhawk Plastic Surgery, Danville, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study subjects were recruited in the medical clinic 01/30/09 through 04/07/09.
Groups:
- Treated and Untreated Thigh: Circumference measurement of RF treated thigh compared to untreated thigh (average of 2.8 treatments and average dosage of 27 kJ) on the same subject
Period: Overall Study
Arm/Group | Treated and Untreated Thigh
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treated And Untreated Thigh: Treated and untreated arms (left and right thighs) on the same subject.
Arm/Group | Treated And Untreated Thigh
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Difference in Circumference of Upper Thigh Between Treated and Untreated Control Arms
Description: Mean difference of change from baseline between two arms: [Treated arm - Untreated arm]
Time Frame: Baseline and 6 months post final treatment
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Upper Thigh
Groups:
- Treated and Untreated Upper Thigh: Treated and untreated arms (left and right thigh) on the same participant
Arm/Group | Treated and Untreated Upper Thigh
Number analyzed (Participants) | 4
Number analyzed (Upper Thigh) | 8
cm | 1.0 (1.7)

2. Secondary Outcome: Subject Satisfaction
Time Frame: Baseline and 6 months post final treatment
Population: Data was not collected due to termination.
Measure: Number; unit: Participants
Arm/Group | Treated and Untreated Thigh
Number analyzed (Participants) | 0

3. Secondary Outcome: Adverse Events
Time Frame: At each visit (treatment and follow-up) or until resolution of AEs
Measure: Number; unit: Event
Units Other Than Participants: Thighs (left or right)
Arm/Group | Treated Thigh
Number analyzed (Participants) | 4
Number analyzed (Thighs (left or right)) | 4
Event
  Erythema | 2
  Edema | 2
  Bruising | 2
  Lumps | 3
  Sensitivity | 3
  Discomfort | 3

4. Primary Outcome: Difference in Circumference of Mid Thigh Between Treated and Untreated Control Arms
Description: Mean difference of change from baseline between two arms: [Treated arm - Untreated arm]
Time Frame: Baseline and 6 months post final treatment
Measure: Mean (Standard Deviation); unit: cm
Units Other Than Participants: Mid Thigh
Groups:
- Treated and Untreated Mid Thigh: Treated and untreated arms (left and right thigh) on the same subject
Arm/Group | Treated and Untreated Mid Thigh
Number analyzed (Participants) | 4
Number analyzed (Mid Thigh) | 8
cm | 0.63 (1.2)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Subjects were assessed and followed up for adverse events at 6 weeks, 3 months and 6 months after the RF treatment.
Arm/Group | Treated Thigh
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Thigh (N=4)
Erythema (Injury, poisoning and procedural complications) | 2 (2)
Edema (Injury, poisoning and procedural complications) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Lumps (Injury, poisoning and procedural complications) | 3 (3)
Sensitivity (Injury, poisoning and procedural complications) | 3 (3)
Discomfort (Injury, poisoning and procedural complications) | 3 (3)

LIMITATIONS AND CAVEATS:
Early termination of the study resulting in analysis of small numbers of subjects, and technical issues with repeatability and reproducibility of circumference measurements leading to termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prepare the study results for publication and presentation in cooperation with Cutera. The Doctor will not publish or present the results of the Study, or speak publicly about it, unless Cutera has first had a reasonable opportunity to review and comment on the contents of the proposed presentation or publication.